CLINICAL TRIAL: NCT06841341
Title: EMG and Ultrasound of Respiratory Muscles and Respective Nerves and to Predict Respiratory Insufficiency in ALS
Brief Title: Electrophysiology and Ultrasound of Respiratory Muscles and Respective Nerves to Predict Respiratory Insufficiency in ALS
Status: Enrolling by invitation | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Other Study IDs: JagiellonianU75
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; electromyography; ultrasound; respiratory muscles; rectus abdominis; sternocleidomastoideus; diaphragm; vagus; accessorius; noninvasive ventilation; respiratory insufficiency
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Respiratory Insufficiency | interventions — Electromyography; Ultrasonography; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ALS: Patients with definite, probable or laboratory-supported probable ALS according to revised el Escorial criteria, who are treated in the neurologic ambulatory of the University Hospital in Cracow (Poland)
  Interventions: Diagnostic Test: electromyography; Diagnostic Test: ultrasonography; Diagnostic Test: Arterial blood gas analysis; Diagnostic Test: slow vital capacity

INTERVENTIONS:
Diagnostic Test: electromyography — electromyography of a set of muscles usually examined during diagnosis of ALS (typically tongue, bilateral deltoid, first dorsal interosseur, abductor pollicis brevis, paraspinals, vastus lateralis, anterior tibialis and additionally bilateral sternocleidomastoideus and rectus abdominis). In each muscle recording in relaxation and in maximal voluntary effort will be done. The presence of signs of acute (fibrillations, sharp waves) and chronic (fasciculations, reduction of the recording of the effort) denervation as well as presence of activity coupled with the rhythm of respiration will be assessed.
Diagnostic Test: ultrasonography — Ultrasonographic measurements include cross-sectional area (CSA) and diameter of bilateral phrenicus, vagus and accessory nerves as well as diameter of diaphragm. The diameter of diaphragm will be measured during normal, quiet respiration as well as at the peak inspiration and expiration.
Diagnostic Test: Arterial blood gas analysis — Assessment of partial oxygen (PaO2) and partial carbondioxide pressure (PaCO2) in arterial blood.
Diagnostic Test: slow vital capacity — Slow vital capacity (SVC) will be measured as the full exhalation done after inspiration which will follow a period of quiet breathing. The test will be performed thrice and the final value will be the average value.

SUMMARY:
Respiratory insufficiency is a common complication in amyotrophic lateral sclerosis (ALS). Survival can be prolonged with noninvasive ventilation (NIV). The goal of this study is to assess the value of electromyography of respiratory muscles as well as the ultrasound of the diaphragm and nerves involved in respiration in predicting the onset of respiratory insufficiency, which may improve the timing of NIV start. The study will recruit 80 patients with definite or probable ALS. Investigations include electromyography of bilateral sternocleidomastoideus and rectus abdominis with assessment of presence of acute and chronic denervation. Ultrasonographic measurements include crosssectional area and diameter of bilateral phrenicus, vagus and accesory nerves as well as diameter of diaphragm. Respiratory insufficiency is asessed with slow vital capacity and partial pressure of arterial oxygen and arterial carbon dioxide. Forthermore, ALS severity is assessed with revised ALS Functional Rating Scale and the symptoms which may reflect respiratory insufficiency even in the absence of dyspnea such as sleepiness, fatigue and depression are assessed with Fatigue Severity Scale, Epworth Sleepiness Scale and Hamilton Depression Rating Scale respectively. SVC and blood gases will be compared between group with and without denervation in investigated muscles. SVC and blood gases will be correlated with corssectional areas and diameters of investigated nerves and diaphragm as well as with the scores obtained in used scales and questionnaires.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare condition with progressing degeneration of upper and lower motor neurons. Main symptoms include muscle weakness, spasticity, atrophy and fasciculations, which lead to gait impairment, dysphagia, dysarthria and loss of hand dexterity. Currently no disease modifying treatment is available and the condition leads to death, usually within three to five years. Respiratory insufficiency is a common complication, especially in later stages of the disease. It results from weakness of respiratory muscles and in some cases also from chronic aspiration pneumonia. It decreases significantly quality of life and may shorten the survival. Not infrequently it is not accompanied by feeling of dyspnea but may be associated with other symptoms like tiredness, sleepiness, and depression. Survival and the quality of life can be improved with noninvasive ventilation (NIV), but the timing of detection of respiratory insufficiency and starting the therapy is crucial to achieve the best possible efficacy. The goal of this study is to assess the value of electromyography of respiratory muscles as well as the ultrasound of the diaphragm and nerves involved in respiration in predicting the onset of respiratory insufficiency. Electromyography is a method commonly used to confirm the diagnosis and neuromuscular ultrasound it is increasingly used along with electromyography to exclude mimics, especially in atypical cases. Investigators hypothesize, including nerves and muscles involved in respiration into electrophysiological and ultrasonographic testing may yield additional benefit of detecting actual or antecedent respiratory failure. The study will recruit 80 patients with definite or probable ALS. Investigations include electromyography of bilateral sternocleidomastoideus and rectus abdominis with assessment of presence of acute and chronic denervation. Ultrasonographic measurements include cross-sectional area and diameter of bilateral phrenicus, vagus and accessory nerves as well as diameter of diaphragm. Respiratory insufficiency is assessed with slow vital capacity and partial pressure of arterial oxygen and arterial carbon dioxide. Furthermore, ALS severity is assessed with revised ALS Functional Rating Scale and the symptoms which may reflect respiratory insufficiency even in the absence of dyspnea such as sleepiness, fatigue and depression are assessed with Fatigue Severity Scale, Epworth Sleepiness Scale and Hamilton Depression Rating Scale respectively. SVC and blood gases will be compared between group with and without denervation in investigated muscles. SVC and blood gases will be correlated with corssectional areas and diameters of investigated nerves and diaphragm as well as with the scores obtained in used scales and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite ALS or probable ALS or clinically probable laboratory supported ALS according to revised El Escorial Criteria [Brooks et al. 2000]

Exclusion Criteria:

* Diagnosis of fronto-temporal dementia
* Significant cognitive or behavioral deficits of other origin, which may disturb the participation in the study
* Medical conditions other than SLA likely to cause respiratory insufficiency, significant changes in the blood gases or SVC
* INR (internal normalized ratio) more than 3 (in the last test performed) in patients with history of coagulation disturbances or intake of oral anticoagulants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the neurologic ambulatory and neurologic clinic of Jagiellonian University Medical College in Cracow.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Relation of denervation in respiratory muscles to PaO2 | Through study completion, an average of 1 year
  Difference in PaO2 between patients with signs of denervation in at least one of the examined respiratory muscles and without signs of denervation.
Relation of denervation in respiratory muscles to PaCO2 | Through study completion, an average of 1 year
  Difference in PaCO2 between patients with signs of denervation in at least one of the examined respiratory muscles and without signs of denervation.
Relation of denervation in respiratory muscles to SVC | Through study completion, an average of 1 year
  Difference in SVC between patients with signs of denervation in at least one of the examined respiratory muscles and without signs of denervation.
Correlation between fatigue and SVC | Through study completion, an average of 1 year
  Correlation between FSS score and SVC.

SECONDARY OUTCOMES:
Correlation of CSA of phrenic nerves with SVC | Through study completion, an average of 1 year
  Correlation of CSA of phrenic nerve (averaged for both sides) with SVC.
Correlation of CSA of accessory nerves with SVC | Through study completion, an average of 1 year
  Correlation of CSA of accessory nerve (averaged for both sides) with SVC.
Correlation of diaphragm diameter with SVC | Through study completion, an average of 1 year
  Correlation of diaphragm diameter (averaged for both sides) with SVC.
Correlation of daytime sleepiness with SVC | Through study completion, an average of 1 year
  Correlation of ESS score with SVC.
Correlation of depression with SVC | Through study completion, an average of 1 year
  Correlation of HDRS score with SVC.

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the scans of collected questionnaires will be available upon request sent to the e-mail: jakub.antczak@uj.edu.pl
Supporting Information: Study Protocol, ICF
Time Frame: After the study is completed for the period of ten years.
Access Criteria: Researchers affiliated in institutions listed on clinicaltrials.gov.

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847